CLINICAL TRIAL: NCT00546637
Title: A Randomized, Double-Blind, Placebo-Controlled Study To Evaluate The Efficacy And Safety Of Fesoterodine As An "Add-On" Therapy In Men With Persistent Overactive Bladder Symptoms Under Monotherapy Of Alpha Blocker For Lower Urinary Tract Symptoms.
Brief Title: Fesoterodine "add-on" Male Overactive Bladder Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer,Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0221009
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Results first posted 2010-11-22 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Overactive Bladder Syndrome
MeSH Terms: interventions — fesoterodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Fesoterodine 4mg or 8mg (Experimental)
  Interventions: Drug: Fesoterodine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fesoterodine — Fesoterodine 4mg or 8mg
  Arms: Fesoterodine 4mg or 8mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of fesoterodine on overactive bladder symptom improvement when added to ongoing alpha blocker treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 40 years and above.
* On a stable and well-tolerated dose of an alpha-blocker prescribed for LUTS for at least 6 weeks prior to screening (Visit 1).
* Persistent symptoms of OAB with urinary frequency >=8 times/24 hours and micturition-related urgency episodes >=3 episode/24 hours.

Exclusion Criteria:

* Contraindication to fesoterodine (antimuscarinics).
* Previous history of acute urinary retention requiring catheterization or severe voiding difficulties in the judgment of the investigator, prior to baseline.
* Unable to follow the study procedures, including completion of self-administered bladder diary and patient reported outcome questionnaires.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 947 (Actual)
Dates: Start 2007-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (123):
- United States (56):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Gilbert, Arizona
  - Pfizer Investigational Site, Litchfield Park, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, San Bernardino, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Jupiter, Florida
  - Pfizer Investigational Site, Orange City, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Dunwoody, Georgia
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Newburgh, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Owings Mills, Maryland
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Flint, Michigan
  - Pfizer Investigational Site, Saint Clair Shores, Michigan
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Utica, Michigan
  - Pfizer Investigational Site, West Bloomfield, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Sewell, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Garden City, New York
  - Pfizer Investigational Site, Kingston, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Poughkeepsie, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Greensboro, North Carolina
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Bethany, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Bala-Cynwyd, Pennsylvania
  - Pfizer Investigational Site, Camp Hill, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Madison, Wisconsin
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Belgium (3):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Leuven
- Brazil (6):
  - Pfizer Investigational Site, Salvador, Estado de Bahia
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Campos do Jordão, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (8):
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Barrie, Ontario
  - Pfizer Investigational Site, North Bay, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Colombia (2):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Bogota, Cundinamarca
- Germany (8):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Hagenow
  - Pfizer Investigational Site, Lauenburg
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Oberursel
  - Pfizer Investigational Site, Wiesbaden
- Greece (3):
  - Pfizer Investigational Site, Ioannina, Ipiros
  - Pfizer Investigational Site, Pátrai
  - Pfizer Investigational Site, Thessaloniki
- India (3):
  - Pfizer Investigational Site, New Delhi, New Delhi
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Lucknow, Uttar Pradesh
- Pfizer Investigational Site, Kuching, Sarawak, Malaysia
- Netherlands (3):
  - Pfizer Investigational Site, Roermond
  - Pfizer Investigational Site, Tilburg
  - Pfizer Investigational Site, Zutphen
- Norway (2):
  - Pfizer Investigational Site, Bodø
  - Pfizer Investigational Site, Oslo
- Philippines (5):
  - Pfizer Investigational Site, Cebu City, Cebu
  - Pfizer Investigational Site, Quezon City, Philippines
  - Pfizer Investigational Site, Bacolod City
  - Pfizer Investigational Site, Makati City
  - Pfizer Investigational Site, Manila
- Poland (5):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Mysłowice
  - Pfizer Investigational Site, Wroclaw
- Pfizer Investigational Site, Singapore, Singapore, Singapore
- Slovakia (5):
  - Pfizer Investigational Site, Bratislava, Slovakia
  - Pfizer Investigational Site, Martin, Slovakia
  - Pfizer Investigational Site, Piešťany, Slovakia
  - Pfizer Investigational Site, Banská Bystrica
  - Pfizer Investigational Site, Skalica
- South Korea (3):
  - Pfizer Investigational Site, Bucheon-si, Gyunggi-do
  - Pfizer Investigational Site, Pusan
  - Pfizer Investigational Site, Seoul
- Spain (3):
  - Pfizer Investigational Site, Martorell, Barcelona
  - Pfizer Investigational Site, Getafe, Madrid
  - Pfizer Investigational Site, Manacor, Palma de Mallorca
- Sweden (4):
  - Pfizer Investigational Site, Borås
  - Pfizer Investigational Site, Jönköping
  - Pfizer Investigational Site, Skövde
  - Pfizer Investigational Site, Stockholm
- Thailand (2):
  - Pfizer Investigational Site, Ratchathewi, Bangkok
  - Pfizer Investigational Site, Amphoe Mueang, Chiang Mai

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221009&StudyName=Fesoterodine%20%22add-on%22%20Male%20Overactive%20Bladder%20Study

RESULTS

PARTICIPANT FLOW:
Groups:
- Fesoterodine 4mg or 8mg: Subjects initially treated with fesoterodine 4 mg once-daily for 4 weeks. At Week 4 visit, the dose of study drug was adjusted through collaborative decision by the investigator and the subject. For those subjects who desired greater symptom improvement and reported acceptable safety and tolerability, fesoterodine dose was increased to 8 mg in a blinded fashion. For the rest of subjects, the dose was maintained at fesoterodine 4 mg.
- Placebo: Subjects were initially treated with placebo once-daily for 4 weeks. At Week 4 visit, the dose of study drug was adjusted through collaborative decision by the investigator and the subject. For those subjects who desired greater symptom improvement and reported acceptable safety and tolerability, the matching placebo for fesoterodine 8 mg tablets was provided to those in the placebo group who choose the dose increase. For the rest of subjects, the dose was maintained at matching placebo.
Period: Overall Study
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Started | 474 | 473
Received Treatment | 471 | 472
Completed | 401 | 424
Not Completed | 73 | 49
Not completed — Adverse Event | 46 | 20
Not completed — Lack of Efficacy | 5 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Other | 10 | 12
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Randomized, but not treated | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fesoterodine 4mg or 8mg | Placebo | Total
Number analyzed (Participants) | 471 | 472 | 943
Age, Customized [Number; unit: participants]
  18 - 44 years | 7 | 9 | 16
  45- 64 years | 211 | 189 | 400
  >=65 years | 253 | 274 | 527
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 471 | 472 | 943

OUTCOME MEASURES:

1. Primary Outcome: Numerical Change From Baseline in Micturition-Related Urgency Episodes Per 24 Hours at Week 12
Description: The mean number of micturition-related urgency episodes per 24 hours was calculated as the total number of micturitions with USS Scale >= 3 divided by the total number of days that diary data was collected at that visit. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline, Week 12
Population: The full analysis set (FAS) included all subjects who took at least one dose of assigned study drug and had at least one baseline or post-baseline efficacy assessment. Only FAS subjects with non-zero micturition-related urgency episodes at Baseline and non-missing change from Baseline to Week 12 (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: number of episodes
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 446 | 451
number of episodes | -3.2 (0.2) | -2.9 (0.2)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; The null hypothesis was that the mean change from Baseline in 24-hour micturition-related urgency was the same at Week 12 for the two treatment groups: fesoterodine + alpha-blocker vs. placebo + alpha-blocker. It was estimated that 900 randomized subjects would have 85% power to detect a mean difference of -0.93(SD = 4.15) between the 2 treatments on the primary endpoint,mean reduction of micturition-related urgency episodes/24hr from Baseline to Week 12,assuming a 10% non-evaluability rate; Test type: Superiority or Other; p = 0.1959, ANCOVA — P-value was based on an ANCOVA model with terms for country, treatment, and baseline value as covariate. No adjustment of p-value was made for multiple comparisons; Mean Difference (Net) = -0.4, 95% CI [-0.9 to 0.2], Standard Error of Mean 0.3 — Mean difference (Net) = Least squares mean

2. Secondary Outcome: Numerical Change From Baseline in Micturition-Related Urgency Episodes Per 24 Hours at Week 4
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: FAS subjects with non-zero baseline and non-missing change from Baseline to Week 4 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: number of episodes
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 445 | 450
number of episodes | -2.3 (0.2) | -1.9 (0.2)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Test type: Superiority or Other; p = 0.0621, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.5, 95% CI [-1.0 to 0.0], Standard Error of Mean 0.2 — Mean difference (net) = Least squares mean

3. Secondary Outcome: Percentage Change From Baseline in Micturition-Related Urgency Episodes Per 24 Hours at Week 4 and 12
Description: Micturition-related urgency episodes per 24 hours were defined as those with USS Scale rating of >= 3 marked for the corresponding micturition in the diary. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. The percentage change at Week 4 or 12 was calculated as:
  100* (Micturition-Related Urgency Episodes at Week 4 or 12 - Baseline)/Baseline
Time Frame: Baseline, Week 4 and 12
Population: FAS subjects with non-zero baseline and non-missing change from Baseline to Week 4 or Week 12 (LOCF) were included in the analysis.
Measure: Median (Full Range); unit: percent change
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 446 | 451
percent change
  Week 4 (n=445, 450) | -30.8 (56.9) [-100.0 to 363.3] | -20.7 (49.1) [-100.0 to 158.8]
  Week 12 (n=446, n=451) | -43.8 (60.8) [-100.0 to 363.6] | -35.7 (58.0) [-100.0 to 600.0]

4. Secondary Outcome: Numerical Change From Baseline in Micturitions Per 24 Hours at Week 4 and 12
Description: All micturitions with USS rating 1 to 5. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. The mean number of micturitions per 24 hours was calculated as the total number of micturitions divided by the total number of diary days collected at that visit. Numeric change of micturitions per 24 hours at Week 4 and 12 relative to Baseline.
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: number of micturitions
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 446 | 452
number of micturitions
  Week 4 (n=445, n=451) | -1.3 (0.1) | -0.8 (0.1)
  Week 12 (n=446, n=452) | -1.9 (0.1) | -1.5 (0.1)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0056, ANCOVA — P-value was based on ANCOVA model with terms for country, treatment, and baseline value as a covariate. No adjustment of p-value was made for multiple comparisons; Mean Difference (Net) = -0.4, 95% CI [-0.8 to -0.1], Standard Error of Mean 0.2 — Mean difference (net) = Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0090, ANCOVA — P-value was based on ANCOVA model with terms for country, treatment, and baseline value as covariate. No adjustment of p-value was made for multiple comparisons; Mean Difference (Net) = -0.4, 95% CI [-0.7 to -0.1], Standard Error of Mean 0.2 — Mean difference (net) = Least squares mean

5. Secondary Outcome: Percentage Change From Baseline in Micturitions Per 24 Hours at Week 4 and 12
Description: All micturitions with USS rating 1 to 5. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. The percentage change at Week 4 or 12 was calculated as: 100* (Micturitions at Week 4 or 12 - Baseline)/Baseline
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 3
Measure: Median (Full Range); unit: percent change
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 446 | 452
percent change
  Week 4 (n=445, n=451) | -12.0 (18.8) [-71.6 to 96.2] | -7.3 (18.9) [-53.7 to 66.7]
  Week 12 (n=446, n=452) | -14.9 (19.3) [-81.8 to 96.2] | -12.5 (19.2) [-58.3 to 51.4]
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0012, Ranked ANCOVA — P-value was based on a ranked ANCOVA model with terms for country, treatment, and ranked baseline value as a covariate. No adjustment of p-value was made for multiple comparisons; Treatment comparisons were performed only if the corresponding numerical change from Baseline at the same visit was statistically significant
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0027, Ranked ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]

6. Secondary Outcome: Numerical Change From Baseline in Nocturnal Micturitions Per 24 Hours at Week 4 and 12
Description: Nocturnal micturitions were defined as micturitions with USS rating 1-5 that occurred between the time the subject went to bed and the time he or she arose to start the next day. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. The mean number of nocturnal micturitions per 24 hours was calculated as the total number of nocturnal micturitions divided by the total number of diary days collected at that visit.
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: number of micturitions
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 439 | 442
number of micturitions
  Week 4 (n=438, n=441) | -0.4 (0.1) | -0.3 (1.0)
  Week 12 (n=439, n=442) | -0.6 (0.1) | -0.5 (0.1)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.1112, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -0.1, 95% CI [-0.2 to 0.0], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0855, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -0.1, 95% CI [-0.3 to 0.0], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean

7. Secondary Outcome: Percentage Change From Baseline in Nocturnal Micturitions Per 24 Hours at Week 4 and 12
Description: Nocturnal micturitions were defined as micturitions with USS rating 1-5 that occurred between the time the subject went to bed and the time he or she arose to start the next day. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. The percentage change at Week 4 or 12 was calculated as: 100* (Nocturnal micturitions at Week 4 or 12 - Baseline)/Baseline
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 3
Measure: Median (Full Range); unit: percent change
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 439 | 442
percent change
  Week 4 (n=438, n=441) | -16.7 (60.4) [-100.0 to 700] | -11.1 (44.8) [-100.0 to 300.0]
  Week 12 (n=439, n=442) | -25.0 (66.1) [-100.0 to 600.0] | -16.7 (58.2) [-100.0 to 700.0]

8. Secondary Outcome: Numerical Change From Baseline in Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 4 and 12
Description: UUI episodes were defined as those micturitions with USS rating of 5 in the diary in subjects with UUI at baseline. USS rating 5: Unable to hold; leak urine.
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 3
Measure: Median (Full Range); unit: number of episodes
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 103 | 104
number of episodes
  Week 4 (n=103, n=104) | -0.3 (1.9) [-11.3 to 5.7] | -0.7 (1.7) [-6.7 to 9.7]
  Week 12 (n=103, n=104) | -0.7 (2.3) [-16.7 to 5.7] | -0.7 (1.4) [-6.7 to 4.0]
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.3847, Van Elteren's Test — P-value was based on Van Elteren's Test adjusted by baseline quartiles. No adjustment of p-value was made for multiple comparisons; Mean Difference (Net) = 0.0 — Median difference was estimated using Hodges-Lehmann estimate of the location shift between the two groups
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.4449, Van Elteren's Test — [p-value comment as in outcome 8, analysis 1]; Median Difference (Net) = 0.0 — Median difference was estimated using Hodges-Lehmann estimate of the location shift between the two groups

9. Secondary Outcome: Percentage Change From Baseline in UUI Episodes Per 24 Hours at Week 4 and 12
Description: UUI episodes are defined as those micturitions with a USS rating of 5 in the bladder diary in subjects with UUI at baseline. USS rating 5: Unable to hold; leak urine. The percentage change at Week 4 or 12 was calculated as: 100* (UUI Episodes at Week 4 or 12 - Baseline)/Baseline
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 3
Measure: Median (Full Range); unit: percent change
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 103 | 104
percent change
  Week 4 (n=103, n=104) | -100.0 (85.3) [-100.0 to 425.0] | -100.0 (136.7) [-100.0 to 966.7]
  Week 12 (n=103, n=104) | -100.0 (77.2) [-100.0 to 425.0] | -100.0 (79.0) [-100.0 to 300.0]

10. Secondary Outcome: Numerical Change From Baseline in Severe Micturition-Related Urgency Episodes Per 24 Hours at Week 4 and 12
Description: Severe micturition related urgency episodes were defined as those micturitions with USS rating >=4 marked for the corresponding micturition in the diary. USS: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 3
Measure: Median (Full Range); unit: number of episodes
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 311 | 340
number of episodes
  Week 4 (n=310, n=339) | -1.0 (2.7) [-13.0 to 10.7] | -1.0 (2.6) [-11.0 to 13.7]
  Week 12 (n=311, n=340) | -1.3 (3.1) [-18.0 to 10.7] | -1.0 (2.8) [-16.7 to 9.0]
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0062, Van Elteren's Test — [p-value comment as in outcome 8, analysis 1]; Median Difference (Net) = -0.33 — Median difference was based on Hodges-Lehmann estimate of the location shift between the two groups
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0825, Van Elteren's Test — [p-value comment as in outcome 8, analysis 1]; Median Difference (Net) = 0.00 — Median difference was based on Hodges-Lehmann estimate of the location shift between the two groups

11. Secondary Outcome: Percentage Change From Baseline in Severe Micturition-Related Urgency Episodes Per 24 Hours at Week 4 and 12
Description: Severe micturition-related urgency episodes are defined as those with a USS rating ≥4 marked for the corresponding micturition in the bladder diary. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. The percentage change at Week 4 or 12 was calculated as: 100* (Severe Micturition-Related Urgency Episodes at Week 4 or 12 - Baseline)/Baseline
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 3
Measure: Median (Full Range); unit: percent change
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 311 | 340
percent change
  Week 4 (n=310, n=339) | -78.6 (79.4) [-100.0 to 500] | -60.0 (130.7) [-100.0 to 1366.7]
  Week 12 (n=311, n=340) | -100.0 (100.7) [-100.0 to 600.0] | -88.4 (90.1) [-100.0 to 600.0]
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0025, Ranked ANCOVA — P-value for median was based on a ranked ANCOVA model with terms for country, treatment, and ranked baseline value as a covariate. No adjustment of p-value was made for multiple comparisons; [statistical method as in outcome 5, analysis 1]

12. Secondary Outcome: Numerical Change From Baseline in Nocturnal Micturition-Related Urgency Episodes Per 24 Hours at Week 4 and 12
Description: Nocturnal micturition-related urgency episodes were defined as micturition-related urgency episodes with USS ratings 3-5 that occurred between the time the subject went to bed and the time he or she arose to start the next day. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: number of episodes
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 425 | 434
number of episodes
  Week 4 (n= 424, n=433) | -0.7 (0.1) | -0.6 (0.1)
  Week 12 (n=425, n=434) | -0.9 (0.1) | -0.9 (0.1)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.1748, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -0.1, 95% CI [-0.3 to 0.0], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.6572, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 0.0, 95% CI [-0.1 to 0.2], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean

13. Secondary Outcome: Percentage Change From Baseline in Nocturnal Micturition-Related Urgency Episodes Per 24 Hours at Week 4 and 12
Description: Nocturnal micturition-related urgency episodes were defined as micturition-related urgency episodes with USS ratings 3-5 that occurred between the time the subject went to bed and the time he or she arose to start the next day. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. The percentage change at Week 4 or 12 was calculated as: 100* (Nocturnal Micturition-Related Urgency Episodes at Week 4 or 12 - Baseline)/Baseline
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 3
Measure: Median (Full Range); unit: percent change
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 425 | 434
percent change
  Week 4 (n=424, n=433) | -33.3 (87.1) [-100.0 to 800.0] | -25.0 (68.9) [-100.0 to 400.0]
  Week 12 (n=425, n=434) | -50.0 (104.2) [-100.0 to 800.0] | -40.0 (70.4) [-100.0 to 400.0]

14. Secondary Outcome: Numerical Change From Baseline in Urinary Sensation Scale (USS) Sum Rating Per 24 Hours at Week 4 and 12
Description: The USS sum rating was defined as the total of USS ratings recorded for all micturitions over the course of a day in the bladder diary. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. USS Sum rating per 24 hours was calculated as the mean rating scores on the USS multiplied by the mean number of micturitions per 24 hours at that visit.
Time Frame: Baseline, Week 4 and 12
Population: FAS subjects with non-missing change from Baseline (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: USS Sum rating per 24 hours
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 446 | 452
USS Sum rating per 24 hours
  Week 4 (n=445, n=451) | -6.4 (0.5) | -4.7 (0.5)
  Week 12 (n=446, n=452) | -8.9 (0.6) | -7.8 (0.6)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0051, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -1.7, 95% CI [-2.9 to -0.5], Standard Error of Mean 0.6 — Mean difference (net) = Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.1231, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -1.0, 95% CI [-2.3 to 0.3], Standard Error of Mean 0.7 — Mean difference (net) = Least squares mean

15. Secondary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) Total Score (Sum Question 1 [Q1] to Q7) Per 24 Hours at Week 4 and 12
Description: The IPSS Total Score is obtained by combining the scores of the responses to 1 though 7 component questions. Each question is scored from 0-5 for an IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
Time Frame: Baseline, Week 4 and 12
Population: FAS subjects with non-missing change from Baseline to Week 4 or Week 12 (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 454 | 456
scores on a scale
  Week 4 (n=453, n=454) | -3.4 (0.3) | -3.1 (0.3)
  Week 12 (n=454, n=456) | -4.4 (0.3) | -4.4 (0.3)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.3579, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.3, 95% CI [-1.0 to 0.4], Standard Error of Mean 0.4 — Mean difference (net) = Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.9274, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.0, 95% CI [-0.8 to 0.7], Standard Error of Mean 0.4 — Mean difference (net) = Least squares mean

16. Secondary Outcome: Change From Baseline in IPSS Storage Domain (Sum Q2, Q4, and Q7) Per 24 Hours at Week 4 and 12
Description: The IPSS Total Score is obtained by combining the scores of the responses to 1 though 7 component questions. Each question is scored from 0-5. Total IPSS range = 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Sum of Q2, Q4, and Q7 range = 0-15 points.
Time Frame: Baseline, Week 4 and 12
Population: FAS subjects with non-missing change from Baseline to Week 4 or Week 12 (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 456 | 458
scores on scale
  Week 4 (n=456, n=457) | -1.8 (0.1) | -1.4 (0.1)
  Week 12 (n=456, n=458) | -2.4 (0.2) | -2.1 (0.2)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0223, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Net) = -0.4, 95% CI [-0.7 to -0.1], Standard Error of Mean 0.2 — Mean difference (net) = Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.1744, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Net) = -0.3, 95% CI [-0.6 to 0.1], Standard Error of Mean 0.2 — Mean difference (net) = Least squares mean

17. Secondary Outcome: Change From Baseline in IPSS Voiding Domain (Sum Q1, Q3, Q5, and Q6) Per 24 Hours at Week 4 and 12
Description: The IPSS Total Score is obtained by combining the scores of the responses to 1 though 7 component questions. Each question is scored from 0-5. Total IPSS range = 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Sum of Q1, Q3, Q5, and Q6 range = 0-20 points.
Time Frame: Baseline, Week 4 and 12
Population: FAS subjects with non-missing change from Baseline to Week 4 or Week 12 (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 455 | 457
scores on scale
  Week 4 (n=454, n=455) | -1.6 (0.2) | -1.7 (0.2)
  Week 12 (n=455, n=457) | -2.1 (0.2) | -2.3 (0.2)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.7564, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Net) = 0.1, 95% CI [-0.4 to 0.5], Standard Error of Mean 0.2 — Mean difference (net) = Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.4010, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Net) = 0.2, 95% CI [-0.3 to 0.7], Standard Error of Mean 0.2 — Mean difference (net) = Least squares mean

18. Secondary Outcome: Change From Baseline in IPSS Quality of Life (QoL) Score (Q8) Per 24 Hours at Week 4 and 12
Description: The IPSS Total Score is obtained by combining the scores of the responses to 1 though 7 component questions. Each question is scored from 0-5. Total IPSS range = 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Score of Q8 range = 0-5 points.
Time Frame: Baseline, Week 4 and 12
Population: FAS subjects with non-missing change from Baseline to Week 4 or Week 12 (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 455 | 457
scores on scale
  Week 4 (n=455, n=455) | -0.6 (0.1) | -0.5 (0.1)
  Week 12 (n=455, 457) | -1.0 (0.1) | -1.0 (0.1)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.1472, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -0.1, 95% CI [-0.2 to 0.0], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.5839, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -0.0, 95% CI [-0.2 to 0.1], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean

19. Secondary Outcome: Change From Baseline in IPSS Individual Item Scores (Q1, Q2, Q3, Q4, Q5, Q6, and Q7) Per 24 Hours at Week 4
Description: The IPSS Total Score is obtained by combining the scores of the responses to 1 though 7 component questions. Each question is scored from 0-5. Total IPSS range = 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
Time Frame: Baseline, Week 4
Population: FAS subjects with non-missing change from Baseline to Week 4 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 445 | 451
scores on scale
  Q1 (sensation of not emptying bladder?) | -0.6 (0.1) | -0.6 (0.1)
  Q2 (urinate less than two hours after urination?) | -0.8 (0.1) | -0.5 (0.1)
  Q3 (stop and start several times during urination? | -0.4 (0.1) | -0.4 (0.1)
  Q4 (difficulty postponing urination?) | -0.7 (0.1) | -0.6 (0.1)
  Q5 (weak urinary stream?) | -0.5 (0.1) | -0.4 (0.1)
  Q6 (strain to begin urination?) | -0.2 (0.1) | -0.3 (0.1)
  Q7 (urinate at night?) | -0.3 (0.1) | -0.3 (0.1)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4 Q1; Test type: Superiority or Other; p = 0.6621, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 0.0, 95% CI [-0.1 to 0.2], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4 Q2; Test type: Superiority or Other; p < .0001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -0.3, 95% CI [-0.5 to -0.2], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 3: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4 Q3; Test type: Superiority or Other; p = 0.3242, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 0.1, 95% CI [-0.1 to 0.2], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 4: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4 Q4; Test type: Superiority or Other; p = 0.1604, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -0.1, 95% CI [-0.3 to 0.0], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 5: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4 Q5; Test type: Superiority or Other; p = 0.4102, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -0.1, 95% CI [-0.2 to 0.1], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 6: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4 Q6; Test type: Superiority or Other; p = 0.3079, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 0.1, 95% CI [-0.1 to 0.2], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 7: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4 Q7; Test type: Superiority or Other; p = 0.4066, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean

20. Secondary Outcome: Change From Baseline in IPSS Individual Item Scores (Q1, Q2,Q3, Q4, Q5, Q6, and Q7) Per 24 Hours at Week 12
Description: as for outcome 15
Time Frame: Baseline, Week 12
Population: FAS subjects with non-missing change from Baseline to Week 12 (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 445 | 451
scores on scale
  Q1 (sensation of not emptying bladder?) | -0.7 (0.1) | -0.8 (0.1)
  Q2 (urinate less than two hours after urination?) | -0.9 (0.1) | -0.8 (0.1)
  Q3 (stop and start several times during urination? | -0.5 (0.1) | -0.6 (0.1)
  Q4 (difficulty postponing urination?) | -0.9 (0.1) | -0.8 (0.1)
  Q5 (weak urinary stream?) | -0.6 (0.1) | -0.6 (0.1)
  Q6 (strain to begin urination?) | -0.3 (0.1) | -0.3 (0.1)
  Q7 (urinate at night?) | -0.5 (0.1) | -0.6 (0.1)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12 Q1; Test type: Superiority or Other; p = 0.1595, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 0.1, 95% CI [-0.0 to 0.3], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12 Q2; Test type: Superiority or Other; p = 0.0614, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -0.2, 95% CI [-0.3 to 0.0], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 3: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12 Q3; Test type: Superiority or Other; p = 0.2032, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 0.1, 95% CI [-0.1 to 0.3], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 4: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12 Q4; Test type: Superiority or Other; p = 0.0631, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -0.2, 95% CI [-0.3 to 0.0], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 5: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12 Q5; Test type: Superiority or Other; p = 0.9706, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -0.0, 95% CI [-0.2 to 0.2], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 6: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12 Q6; Test type: Superiority or Other; p = 0.8058, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 0.0, 95% CI [-0.1 to 0.2], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean
Statistical Analysis 7: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12 Q7; Test type: Superiority or Other; p = 0.3302, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.1 — Mean difference (net) = Least squares mean

21. Secondary Outcome: Number of Participants With Change From Baseline in Patient Perception of Bladder Condition (PPBC) Per 24 Hours at Week 4
Description: PPBC: self-administered, single-item, validated questionnaire. Rated on a 6-point scale: subject was asked: "Which of the following statements describes your bladder condition best at the moment?" 1=no problems at all; 2=some very minor problems; 3=some minor problems; 4=some moderate problems; 5=severe problems; 6=many severe problems. A post-baseline vs baseline variable with ordinal values was derived: 1=Deterioration=Difference in scores was positive; 2=No Change=Difference in scores was 0; 3=Minor Improvement=Difference in scores was -1; 4=Major Improvement=Difference in scores was ≤ 2.
Time Frame: Baseline, Week 4
Population: FAS subjects with non-missing Baseline and Week 4 values.
Measure: Number; unit: participants
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 459 | 457
participants
  Major Improvement | 83 | 63
  Minor Improvement | 171 | 160
  No Change | 180 | 212
  Deterioration | 25 | 22
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Test type: Superiority or Other; p = 0.1136, Cochran-Mantel-Haenszel — P-value was obtained from a Cochran-Mantel-Haenszel test with modified ridit scoring, stratified by center. No adjustment of p-value was made for multiple comparisons

22. Secondary Outcome: Number of Participants With Change From Baseline in PPBC Per 24 Hours at Week 12
Description: as for outcome 21
Time Frame: Baseline, Week 12
Population: FAS subjects with non-missing Baseline and Week 12 values (LOCF).
Measure: Number; unit: participants
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 459 | 459
participants
  Major Improvement | 124 | 130
  Minor Improvement | 166 | 138
  No Change | 148 | 170
  Deterioration | 21 | 21
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Test type: Superiority or Other; p = 0.5775, Cochran-Mantel-Haenszel — [p-value comment as in outcome 21, analysis 1]

23. Secondary Outcome: Number of Participants With Change From Baseline in Urgency Perception Scale (UPS) Per 24 Hours at Week 4
Description: Number of participants in 3-point category: improvement [>=1-point improvement]; no change; deterioration [>=1-point decrease], based on UPS score (rated on 3-point scale: 1=not able to hold urine; 3=able to finish what I am doing). Score change calculated as score at observation minus score at baseline; re-scaled to 3-point categorical variables.
Time Frame: Baseline, Week 4
Population: FAS subjects with non-missing Baseline and Week 4 values.
Measure: Number; unit: participants
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 458 | 458
participants
  Improvement | 111 | 98
  No Change | 306 | 326
  Deterioration | 41 | 34
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Test type: Superiority or Other; p = 0.7433, Cochran-Mantel-Haenszel — [p-value comment as in outcome 21, analysis 1]

24. Secondary Outcome: Number of Participants With Change From Baseline in Change From Baseline in UPS Per 24 Hours at Week 12.
Description: as for outcome 23
Time Frame: Baseline, Week 12
Population: FAS subjects with non-missing Baseline and Week 12 values (LOCF).
Measure: Number; unit: participants
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 459 | 459
participants
  Improvement | 132 | 129
  No Change | 290 | 299
  Deterioration | 37 | 31
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Test type: Superiority or Other; p = 0.9402, Cochran-Mantel-Haenszel — [p-value comment as in outcome 21, analysis 1]

25. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire (OAB-q) Per 24 Hours at Week 4 and 12
Description: OAB-q is a self-administered, 33-item, validated questionnaire that assesses how much the subject has been bothered by selected bladder symptoms during the previous week. Each item rated by subject on Likert scale 1 (least symptom bother) to 6 (most symptom bother). Raw scores were transformed to a score from 0-100. Once transformed, higher scores represent less favorable outcome.
Time Frame: Baseline, Week 4 and 12
Population: FAS subjects with non-missing change from Baseline to Week 4 or Week 12 (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 459 | 459
scores on scale
  Week 4 (n=459, n=458) | -11.6 (0.8) | -8.9 (0.8)
  Week 12 (n=459, n=459) | -15.2 (0.9) | -12.4 (0.9)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0040, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -2.7, 95% CI [-4.5 to -0.9], Standard Error of Mean 0.9 — Mean difference (net) = Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0068, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = -2.8, 95% CI [-4.8 to -0.8], Standard Error of Mean 1.0 — Mean difference (net) = Least squares mean

26. Secondary Outcome: Change From Baseline in Total Score of Each Health Related Quality of Life (HRQL) Domain of OAB-q at Week 4 and 12
Description: HRQL domain and total raw score derived as sum of scores (6-point scale: 1 = not at all/none of the time; 6 = a very great deal/all of the time). Transformed score range 0 to 100 (Total HRQL or domain)=[(Highest possible raw score-Actual total raw score)/Raw score range]x100. Higher transformed scores indicative of better HRQL. Positive change in HRQL scores indicates improvement. Change: score at observation minus score at baseline.
Time Frame: Baseline, Week 4 and 12
Population: FAS subjects with non-missing change from Baseline to Week 4 or Week 12 (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 459 | 459
scores on scale
  Week 4 (n=459, n=458) | 8.7 (0.8) | 6.9 (0.8)
  Week 12 (n=459, n=459) | 11.5 (0.8) | 10.0 (0.9)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0412, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 1.9, 95% CI [0.1 to 3.6], Standard Error of Mean 0.9 — Mean Difference (net)= Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.1373, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 1.5, 95% CI [-0.5 to 3.4], Standard Error of Mean 1.0 — Mean Difference (net)= Least squares mean

27. Secondary Outcome: Change From Baseline in Score of Each Health Related Quality of Life (HRQL) Domain of OAB-q at Week 4 and 12 (OAB-q Concern Domain)
Description: The HRQL concern domain; range was 0-100. The transformed score for HRQL was calculated based on the following formula: Transformed score (HRQL) = [(Highest possible score - Actual raw score)/ Range]*100, where range was the raw score range. Positive change in HRQL Score indicates improvement.
Time Frame: Baseline, Week 4 and 12
Population: FAS subjects with non-missing change from Baseline to Week 4 or Week 12 (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 459 | 459
scores on scale
  Week 4 (n=459, n=458) | 9.7 (0.9) | 8.0 (0.9)
  Week 12 (n=459, n=459) | 12.4 (0.9) | 11.1 (0.9)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0941, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 1.7, 95% CI [-0.3 to 3.8], Standard Error of Mean 1.0 — Mean Difference (net) = Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.2273, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 1.3, 95% CI [-0.8 to 3.4], Standard Error of Mean 1.1 — Mean Difference (net) = Least squares mean

28. Secondary Outcome: Change From Baseline in Score of Each Health Related Quality of Life (HRQL) Domain of OAB-q at Week 4 and 12 (OAB-q Coping Domain)
Description: The HRQL coping domain; range was 0-100. The transformed score for HRQL was calculated based on the following formula: Transformed score (HRQL) = [(Highest possible score - Actual raw score)/ Range]*100, where range was the raw score range. Positive change in HRQL Score indicates improvement.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS subjects with non-missing change from Baseline to Week 4 or Week 12 (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 459 | 459
scores on a scale
  Week 4 (n=459, n=458) | 9.6 (0.9) | 7.5 (0.9)
  Week 12 (n=459, n=459) | 12.5 (1.0) | 10.6 (1.0)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0507, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 2.1, 95% CI [-0.0 to 4.3], Standard Error of Mean 1.1 — Mean Difference (net)= Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.1136, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 1.9, 95% CI [-0.4 to 4.1], Standard Error of Mean 1.2 — Mean Difference (net)= Least squares mean

29. Secondary Outcome: Change From Baseline in Score of Each Health Related Quality of Life (HRQL) Domain of OAB-q at Week 4 and 12 (OAB-q Sleep Domain)
Description: The HRQL sleep domain; range was 0-100. The transformed score for HRQL was calculated based on the following formula: Transformed score (HRQL) = [(Highest possible score - Actual raw score)/ Range]*100, where range was the raw score range. Positive change in HRQL Score indicates improvement.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS subjects with non-missing change from Baseline to Week 4 or Week 12 (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 459 | 459
scores on a scale
  Week 4 (n=459, n=458) | 9.6 (1.0) | 7.6 (1.0)
  Week 12 (n=459, n=459) | 13.8 (1.0) | 11.5 (1.1)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0845, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 1.9, 95% CI [-0.3 to 4.1], Standard Error of Mean 1.1 — Mean Difference (net)= Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0662, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 2.2, 95% CI [-0.2 to 4.6], Standard Error of Mean 1.2 — Mean Difference (net) = Least squares mean

30. Secondary Outcome: Change From Baseline in Score of Each Health Related Quality of Life (HRQL) Domain of OAB-q at Week 4 and 12 (OAB-q Social Interaction Domain)
Description: The HRQL social interaction domain; range was 0-100. The transformed score for HRQL was calculated based on the following formula: Transformed score (HRQL) = [(Highest possible score - Actual raw score)/ Range]*100, where range was the raw score range. Positive change in HRQL Score indicates improvement.
Time Frame: Baseline, Week 4 and Week 12
Population: FAS subjects with non-missing change from Baseline to Week 4 or Week 12 (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 459 | 459
scores on a scale
  Week 4 (n=459, n=458) | 5.2 (0.8) | 3.7 (0.8)
  Week 12 (n=459, n=459) | 6.3 (0.8) | 6.0 (0.8)
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.1085, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 1.4, 95% CI [-0.3 to 3.2], Standard Error of Mean 0.9 — Mean Difference (net) = Least squares mean
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.7685, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Mean Difference (Net) = 0.3, 95% CI [-1.6 to 2.1], Standard Error of Mean 0.9 — Mean Difference (net) = Least squares mean

31. Secondary Outcome: Change From Baseline in Post Void Residual (PVR) Urine Volume Per 24 Hours at Week 4, 8 and 12
Description: Post-void residual volume measurement was measured by an ultrasound at Baseline, and at Weeks 4, 8 and 12.
Time Frame: Baseline, Week 4, 8 and 12
Population: The safety analysis set included all subjects who took at least one dose of study drug. Subjects in the safety analysis set with non missing change from Baseline to Week 4, Week 8 (LOCF), or Week 12 (LOCF) were included in the analysis.
Measure: Median (Full Range); unit: ml
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 454 | 453
ml
  Week 4 | 0.0 [-174.0 to 274.0] | 0.0 [-251.0 to 193.0]
  Week 8 | 0.0 [-180.0 to 275.0] | 0.0 [-180.0 to 255.0]
  Week 12 | 3.5 [-156.0 to 392.0] | 0.0 [-172.0 to 405.0]
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0005, Van Elteren's Test — [p-value comment as in outcome 8, analysis 1]; Median Difference (Net) = 6.00 — Median difference was based on Hodges-Lehmann estimate of the location shift between the two groups
Statistical Analysis 2: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 8; Test type: Superiority or Other; p < .0001, Van Elteren's Test — [p-value comment as in outcome 8, analysis 1]; Median Difference (Net) = 7.00 — Median difference was based on Hodges-Lehmann estimate of the location shift between the two groups
Statistical Analysis 3: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0003, Van Elteren's Test — [p-value comment as in outcome 8, analysis 1]; Median Difference (Net) = 9.00 — Median difference was based on Hodges-Lehmann estimate of the location shift between the two groups

32. Secondary Outcome: Change From Baseline in Maximum Urinary Flow Rate (QMAX) Per 24 Hours at Week 12
Description: Maximum urinary flow rate (Qmax) was recorded at Baseline and Week 12 visit.
Time Frame: Baseline, Week 12
Population: The safety analysis set included all subjects who took at least one dose of study drug. Subjects in the safety analysis set with non missing change from Baseline to Week 12 (LOCF) were included in the analysis.
Measure: Median (Full Range); unit: ml/sec
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 425 | 427
ml/sec | 0.0 [-46.9 to 47.4] | 0.0 [-25.9 to 43.0]
Statistical Analysis 1: Comparison: Fesoterodine 4mg or 8mg vs Placebo; Test type: Superiority or Other; p = 0.2251, Van Elteren's Test — [p-value comment as in outcome 8, analysis 1]; Median Difference (Net) = -0.40 — Median difference was based on Hodges-Lehmann estimate of the location shift between the two groups

33. Secondary Outcome: Number of Participants Reporting Urinary Retention Requiring Catheterization (All Causalities)
Description: Number of participants experiencing serious and non-serious adverse events of acute urinary retention requiring catheterization.
Time Frame: Baseline, Week 12
Population: The safety analysis set included all subjects who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 471 | 472
participants | 1 | 1

34. Secondary Outcome: Number of Participants Experiencing Adverse Events Related to Increased Voiding Difficulty (All Causalities)
Description: Number of participants experiencing serious and non-serious adverse events related to increased voiding difficulty (ie, Dysuria, Urinary retention regardless of catheterization, Urine flow decreased, Residual urine volume, Residual urine volume increased, Residual urine, and Urinary hesitation)
Time Frame: Baseline, Week 12
Population: The safety analysis set included all subjects who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Number analyzed (Participants) | 471 | 472
participants
  Dysuria | 16 | 4
  Urinary retention (Regardless of catheterization) | 11 | 2
  Urine flow decreased | 4 | 0
  Residual urine volume | 1 | 0
  Residual urine volume increased | 1 | 0
  Residual urine | 1 | 0
  Urinary hesitation | 0 | 2

ADVERSE EVENTS:
Arm/Group | Fesoterodine 4mg or 8mg | Placebo
Serious Adverse Events (participants affected / at risk) | 11/471 | 11/472
Other Adverse Events (participants affected / at risk) | 176/471 | 72/472
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine 4mg or 8mg (N=471) | Placebo (N=472)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Genitourinary tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine 4mg or 8mg (N=471) | Placebo (N=472)
Abdominal pain (Gastrointestinal disorders) | 6 | 2
Constipation (Gastrointestinal disorders) | 31 | 10
Diarrhoea (Gastrointestinal disorders) | 9 | 6
Dry mouth (Gastrointestinal disorders) | 100 | 29
Dyspepsia (Gastrointestinal disorders) | 9 | 1
Gastritis (Gastrointestinal disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 6 | 3
Influenza (Infections and infestations) | 6 | 3
Nasopharyngitis (Infections and infestations) | 5 | 2
Sinusitis (Infections and infestations) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 9
Dizziness (Nervous system disorders) | 6 | 8
Headache (Nervous system disorders) | 15 | 8
Insomnia (Psychiatric disorders) | 9 | 5
Dysuria (Renal and urinary disorders) | 15 | 4
Urinary retention (Renal and urinary disorders) | 11 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.